CLINICAL TRIAL: NCT02630056
Title: Validate the Dosimetric Parameters That Correlate With Acute Hematologic Toxicity (HT) in Patients With Rectal Cancer Treated With Neoadjuvant Chemoradiotherapy
Brief Title: Validate the Dosimetric Parameters That Correlate With Acute Hematologic Toxicity (HT) in Patients With Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SASYSU
Record Dates: First submitted 2015-11-27; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-11

CONDITIONS: Rectal Neoplasm
Keywords: radiotherapy hematologic toxicity pelvic bone marrow
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to validate the dosimetric parameters that correlate with acute hematologic toxicity (HT) in patients with rectal cancer treated with neoadjuvant chemoradiotherapy.

DETAILED DESCRIPTION:
The investigators' ongoing retrospective study investigated the clinical and dosimetric parameter (dosimetry of pelvic bone marrow) which relate with acute hematologic toxicity in patient with rectal cancer treated with neoadjuvant chemoradiotherapy. In order to validate the dosimetric limitation of pelvic bone marrow in decreasing the intensity of HT, the investigators want to conduct a study to observe the acute HT without assigning any specific interventions to the subjects of the study, who will receive the standard treatment according to the multidisciplinary team's (MDT) decision and patient choice. Therefore, this study's type is observational.

ELIGIBILITY:
Inclusion Criteria:

* rectal cancer
* receive neoadjuvant chemoradiotherapy

Exclusion Criteria:

* hematological system disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both gender is OK and there is no limitation for age.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the grade of acute hematologic toxicity | 5-6 weeks
  Hematologic Adverse Events That Are Related to Pelvic Bone Marrow Irradiation